CLINICAL TRIAL: NCT05834751
Title: Clinical Study on the Effectiveness and Safety of Pegylated Recombinant Human Granulocyte Stimulating Factor Injection and PEG-rhG-CSF in Mobilizing Autologous Hematopoietic Stem Cells in Lymphoma.
Brief Title: the Efficacy and Safety of PEG-rhG-CSF in Mobilizing Autologous Hematopoietic Stem Cells in Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ou Bai, MD/PHD (Other)
Responsible Party: Sponsor-Investigator, Ou Bai, MD/PHD, Director, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-JYL-PBSCT-03A
Record Dates: First submitted 2023-04-06; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): PEG-rhG-CSF
  Interventions: Drug: PEG-rhG-CSF
- control group (Active Comparator): rhG-CSF
  Interventions: Drug: RhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — 48-72 hours after chemotherapy,9 mg of PEG-rhG-CSF was injected subcutaneously for mobilization
  Other Names: pegfilgrastim
  Arms: experimental group
Drug: RhG-CSF — After clinical evaluation, rhG-CSF was given 10μ g/kg/d for mobilization until the stem cell collection was completed.
  Other Names: filgrastim
  Arms: control group

SUMMARY:
A single center, non-inferiority, two-way cohort clinical study to evaluate the efficacy and safety of pegylated recombinant human granulocyte stimulating factor injection in the mobilization of autologous hematopoietic stem cells in lymphoma.

DETAILED DESCRIPTION:
The objective was to to evaluate the efficacy and safety of pegylated recombinant human granulocyte stimulating factor injection in the mobilization of autologous hematopoietic stem cells in lymphoma.

lymphoma patients who need to be prepared for autologous hematopoietic stem cell transplantation; KPS score ≥70; Ccr≥ 50 mL/min, TBIL< 25.65 umol/L, ALT and AST < 2 times the upper limit of normal value;

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, regardless of gender;
2. lymphoma patients who need to be prepared for autologous hematopoietic stem cell transplantation;
3. KPS score ≥70;
4. Ccr≥ 50 mL/min, TBIL< 25.65 umol/L, ALT and AST < 2 times the upper limit of normal value;
5. ANC ≥ 1.5×109/L，PLT ≥ 80×109/L，Hb ≥ 75g/L，WBC ≥ 3.0×109/L；
6. Patients can tolerate chemotherapy；
7. No active infection before chemotherapy;
8. The retrospective enrolled subjects are exempted from informed consent for data collection, and the prospective enrolled subjects voluntarily participate in this experiment and sign the informed consent form;
9. The researcher thinks that the subjects can benefit.

Exclusion Criteria:

1. Patients with megaspleen (when inhaling deeply, the spleen exceeds the right umbilicus and/or below the umbilical level);
2. Those who have received mobilization and transplantation of allogeneic or autologous hematopoietic stem cells before;
3. Subjects who have evidence of serious or uncontrollable systemic diseases (such as unstable or irreparable respiratory, heart, liver or kidney diseases) according to the researcher's judgment;
4. severe mental or nervous system diseases;
5. Those who are allergic to PEG-rhG-CSF, rhG-CSF and any active ingredients or auxiliary materials of other preparations expressed by Escherichia coli, or have a clear history of protein drug allergy, specific allergic reaction (asthma, rheumatism, eczema dermatitis) or have had other serious allergic reactions;
6. pregnant or lactating female patients; Women of childbearing age refuse to accept contraceptive measures; Those who plan to become pregnant during the study period;
7. The researcher judges other subjects who are not suitable to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Mobilization success rate | 48 months
  Accumulate CD34+cells ≥ 2×106/kg for 3 times or less

SECONDARY OUTCOMES:
White blood cell trough and peak | 30 days
  The treatment period is from the beginning of chemotherapy to the end of collection, the trough value is recorded at the beginning of chemotherapy, and the peak value is recorded after PEG-rhG-CSF is applied
Speed of recovery | 30 days
  The number of days when the leucocyte trough rose to the peak
Time of highest point of CD34+ cells | 30 days
  Time of highest point of CD34+ cells
Single acquisition volume | 30 days
  Single acquisition volume
Acquisition times | 30 days
  Acquisition times
Administration times of rhG-CSF | 30 days
  Administration times of rhG-CSF

CONTACTS AND LOCATIONS:
Overall Officials: Ou Bai, doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang B, Cao L, Li J, Zhao Y, Li J, Wen Y, Yan P, Guo W, Bai O. Polyethylene glycol-conjugated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF) primary prophylaxis significantly reduces the duration of neutropenia in non-Hodgkin's lymphoma patients treated with chemotherapy: a randomised trial (NCT05834751). Transl Cancer Res. 2025 Dec 31;14(12):8990-9001. doi: 10.21037/tcr-2025-1-2613. Epub 2025 Dec 29. PMID 41510127